CLINICAL TRIAL: NCT00250705
Title: Open Label Trial of Aripiprazole in the Treatment of CD in Adolescents
Brief Title: Trial of Aripiprazole in the Treatment of CD in Adolescents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Samuel Kuperman, M.D., Professor, University of Iowa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200306035
Record Dates: First submitted 2005-11-04; First posted 2005-11-08 (Estimated); Results first posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Conduct Disorder
Keywords: Aripiprazole
MeSH Terms: conditions — Conduct Disorder | interventions — Aripiprazole

STUDY DESIGN:
Intervention Model Description: open label trial
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adolescent Conduct Disorder Males (Other): All subjects were male and had a diagnosis of conduct disorder. All subjects were offered treatment with aripiprazole.
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole — The initial dose depending on the weight of the patient will be as follows: < 25 kg = 1 mg/d; 25-50 kg = 2 mg/d; 50-70 kg = 5 mg/d; > 70 kg = 10 mg/d (Data on File, 2003, Bristol-Myers Squibb). Thereafter the dose will be flexible based on response and tolerance for the duration of the 6 week study. All subjects initially received either a 5 or 10 mg/d (7.0 ± 2.6 mg/d) dose of aripiprazole. Thereafter the dose was individualized based on response and tolerance. Maximum dose was 20 mg.
  Other Names: Abilify

SUMMARY:
The proposed study will be a 6-week open label study evaluating aripiprazole in the treatment of 12 male post-pubertal adolescents (13-17 years, Tanner Stage 4) diagnosed with conduct disorder. The initial dose depending on the weight of the patient will be as follows: < 25 kg = 1 mg/d; 25-50 kg = 2 mg/d; 50-70 kg = 5 mg/d; > 70 kg = 10 mg/d (Data on File, 2003, Bristol-Myers Squibb). For the first two weeks of the study, the dose will be flexible based on response and tolerance and thereafter will remain fixed.

DETAILED DESCRIPTION:
The use of atypical antipsychotics in children began in 1992 with several small case series with clozapine. Since that time, five other atypical agents, risperidone, olanzapine, quetiapine, ziprasidone and aripiprazole have been introduced into the US market. The newer atypical agents are not associated with agranulocytosis that has limited the usefulness of clozapine. Among the atypical antipsychotics, risperidone has remained the most extensively studied in children and adolescents, for a variety of problems, including Tourette's disorder, conduct disorder, schizophrenia, aggression, and pervasive development disorder. Risperidone has been shown to be an effective treatment in many of these disorders. However, weight gain, hyperprolactinemia, and extrapyramidal symptoms (EPS) are troublesome adverse effects more commonly associated with risperidone such that the drug's utility in this aged patient population is limited. We expect that the utility of aripiprazole in treating the pediatric population will not be limited by adverse effects like the other atypical antipsychotics.

ELIGIBILITY:
Inclusion Criteria:

* Male post-pubertal adolescents (13-17 years, Tanner Stage 4) diagnosed with conduct disorder.

Exclusion Criteria:

* Clinically significant laboratory and/or ECG abnormalities
* Pre-existing health conditions that would compromise patient safety
* Mental retardation
* Previous use of aripiprazole
* Active psychosis

Ages: 13 Years to 17 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2004-11-17 (Actual); Primary Completion 2009-03-23 (Actual); Study Completion 2009-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Kuperman, M.D., Principal Investigator — University of Iowa
Locations (1):
- The University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kuperman S, Calarge C, Kolar A, Holman T, Barnett M, Perry P. An open-label trial of aripiprazole in the treatment of aggression in male adolescents diagnosed with conduct disorder. Ann Clin Psychiatry. 2011 Nov;23(4):270-6. PMID 22073384

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited through the child psychiatric clinic after being identified as diagnosed with DSM 4 conduct disorder. Subjects and their parents were approached about participation in the study. Recruitment time was November 2004 through March 2009
Pre-assignment Details: The study was an open label study with no separate treatment groups, i.e., different doses or placebo. All subjects that were enrolled into participation were entered into active treatment.
Groups:
- Aripiprazole Treatment of Conduct Disorde: The study was a 6-week open label study evaluating aripiprazole in the treatment of 12 male post-pubertal adolescents (13-17 years, Tanner Stage 4) diagnosed with conduct disorder (American Psychiatric Association 2000). The initial aripiprazole dose depending on the weight of the patient was: < 25 kg = 1 mg/d; 25-50 kg = 2 mg/d; 50-70 kg = 5 mg/d; > 70 kg = 10 mg/d (Data on File, 2003, Bristol-Myers Squibb). Thereafter the dose was individualized based on the response and tolerance to the drug with a maximum aripiprazole dose of 20 mg/d. Current psychotropic medications were not washed out of the patients at the beginning of the study due to the exploratory stage of use of the drug for the conduct disorder indication.
Period: Overall Study
Arm/Group | Aripiprazole Treatment of Conduct Disorde
Started | 12
Completed | 10
Not Completed | 2
Not completed — Lack of Efficacy | 2

BASELINE CHARACTERISTICS:
Groups:
- Aripiprazole Treatment of Conduct Disorder: The study was a 6-week open label study evaluating aripiprazole in the treatment of 12 male post-pubertal adolescents (13-17 years, Tanner Stage 4) diagnosed with conduct disorder (American Psychiatric Association 2000).
Arm/Group | Aripiprazole Treatment of Conduct Disorder
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.6 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Rating of Aggression Against People and/or Property Scale [Mean (Standard Deviation); unit: scores on a scale] — Rating of Aggression Against People and/or Property Scale (RAAPP) (Kemph et al 1993) is a global rating scale of aggression completed by clinicians. Score given based on following severity scale with subject assigned 1 number: Intolerable behavior-frequently physically attacks others and destroys property (5); Severe-occasionally physically attacks people and destroys property (4); Moderately 21); and No aggressiveness reported (1). A minimum score of 1 is best and a maximum score of 5 is worst. There are no subscale scores. Population: 10 subjects who completed the study with last visit carried forward for two.
  scores on a scale | 3.0 (0.9)
Overt Aggression Scale-Modified (OAS-M) (Kay et al 1988) [Mean (Standard Deviation); unit: weighted scores on a scale] — OAS-M divides aggressions into 4 subtypes: 1) verbal, 2) property, 3) self (autoaggression), and 4) physical. Each subtype has an initial score ranging from 0 (least aggressive) to 4 (most aggressive). The score for each subscale is further weighed (multiplied) by a constant: verbal scale's constant is 1 (max adjusted score of 4); property scale's constant is 2 (max adjusted score 8); self scale's constant is 3 (max adjusted score 12); and physical scale's constant is 4 (max adjusted score of 16). Within a given scale, "0" is the best score and maximum adjusted scale score is worst.
  weighted scores on a scale
    OAS-M, verbal aggression | 2.2 (1.2)
    OAS-M, aggression against property | 4.2 (3.0)
    OAS-M, autoaggression | 0.6 (1.9)
    OAS-M, physical aggression | 4.5 (3.9)
Children's Aggression Scale-Parent Version [Mean (Standard Deviation); unit: units on a scale] — CAS-P is a 33 item scale representing 5 domains of aggression: Items in a domain were computed based on two reference points. The first was based on a 5 point frequency range with "0" being best (never) and "4" (> 10 times being) worst. These same items were then adjusted such that more severe acts would be weighted more heavily compared to less severe aggressive behaviors. Within a domain, 0 was the best score. Worst score for the various aggression domains were: Verbal 26.16, Against Objects and Animals 11.8, Provoked 15.84, Initiated 17.84, and Use of Weapons 13.16
  units on a scale
    Verbal Aggression | 12.9 (4.3)
    Agression Against Objects and Animals | 3.8 (2.2)
    Provoked Aggression | 2.1 (2.2)
    Initiated Aggression | 1.6 (2.0)
    Use of Weapons | 0.4 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Efficacy Measure: Rating of Aggression Against People and/or Property Scale (RAAPP) (Kemph et al 1993)
Description: Rating of Aggression Against People and/or Property Scale (RAAPP) (Kemph et al 1993) is a global rating scale of aggression completed by clinicians. Score given based on following severity scale with subject assigned 1 number: Intolerable behavior-frequently physically attacks others and destroys property (5); Severe-occasionally physically attacks people and destroys property (4); Moderately 21); and No aggressiveness reported (1). A minimum score of 1 is best and a maximum score of 5 is worst. There are no subscale scores.
Time Frame: 6 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Aripiprazole Treatment of Conduct Disorder: The study was a 6-week open label study evaluating aripiprazole in the treatment of 10 male post-pubertal adolescents (13-17 years, Tanner Stage 4) diagnosed with conduct disorder (American Psychiatric Association 2000). The initial aripiprazole dose depending on the weight of the patient was: < 25 kg = 1 mg/d; 25-50 kg = 2 mg/d; 50-70 kg = 5 mg/d; > 70 kg = 10 mg/d (Data on File, 2003, Bristol-Myers Squibb). Thereafter the dose was individualized based on the response and tolerance to the drug with a maximum aripiprazole dose of 20 mg/d. Current psychotropic medications were not washed out of the patients at the beginning of the study due to the exploratory stage of use of the drug for the conduct disorder indication.
Arm/Group | Aripiprazole Treatment of Conduct Disorder
Number analyzed (Participants) | 10
units on a scale | 1.7 (0.8)

2. Primary Outcome: Overt Aggression Scale-Modified (OAS-M)
Description: OAS-M divides aggressions into 4 subtypes: 1) verbal aggression, 2) property aggression, 3) self aggression (autoaggression), and 4) physical aggression. Each subtype has an initial score ranging from 0 (least aggressive) to 4 (most aggressive). The score for each subscale is further weighed (multiplied) by a constant: verbal scale's constant is 1 (max adjusted score of 4); property scale's constant is 2 (max adjusted score 8); self scale's constant is 3 (max adjusted score 12); and physical scale's constant is 4 (max adjusted score of 16). Within a given scale, "0" is the best score and maximum adjusted scale score is worst.
Time Frame: 6 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Adolescent Conduct Disorder Males: All subjects were male and had a diagnosis of conduct disorder. All subjects were offered treatment with aripiprazole.
  Aripiprazole: The initial dose depending on the weight of the patient will be as follows: < 25 kg = 1 mg/d; 25-50 kg = 2 mg/d; 50-70 kg = 5 mg/d; > 70 kg = 10 mg/d (Data on File, 2003, Bristol-Myers Squibb). Thereafter the dose will be flexible based on response and tolerance for the duration of the 6 week study. All subjects initially received either a 5 or 10 mg/d (7.0 ± 2.6 mg/d) dose of aripiprazole. The dose was individualized based on response and tolerance with a maximum of 20 mg per day.
Arm/Group | Adolescent Conduct Disorder Males
Number analyzed (Participants) | 10
units on a scale
  verbal aggression | 1.0 (1.2)
  property aggression | 0.6 (1.9)
  self aggression | 0.6 (1.9)
  physical aggression | 1.6 (3.9)

3. Secondary Outcome: Secondary Outcome Measures Were the Clinical Global Impression-Severity (CGI-S) Scale (NIMH, 1985a).
Description: The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Possible ratings are: 1. Normal, not at all ill; 2. Borderline mentally ill, 3. Mildly ill; 4. Moderately ill; 5. Markedly ill; 6. Severely ill; or 7. Among the most extremely ill patients.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aripiprazole Treatment of Conduct Disorder
Number analyzed (Participants) | 10
units on a scale | 3.0 (1.5)

4. Primary Outcome: Children's Aggression Scale-Parent Version
Description: CAS-P is a 33 item scale representing 5 domains of aggression: Items in a domain were computed based on two reference points. The first was based on a 5 point frequency range with "0" being best (never) and "4" (> 10 times being) worst. These same items were then adjusted such that more severe acts would be weighted more heavily compared to less severe aggressive behaviors. Within a domain, 0 was the best score. Worst score for the various aggression domains were: Verbal 26.16, Against Objects and Animals 11.8, Provoked 15.84, Initiated 17.84, and Use of Weapons 13.16.
Time Frame: 6 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adolescent Conduct Disorder Males
Number analyzed (Participants) | 10
units on a scale
  Verbal Aggression | 2.7 (2.8)
  Aggression Against Objects and Animals | 0.4 (0.8)
  Provoked Aggression | 1.6 (0.5)
  Initiated Aggression | 0.6 (1.2)
  Aggression with Use of Weapons | 0.1 (0.3)

5. Secondary Outcome: Secondary Outcome Measures Were the Clinical Global Impression--Improvement (CGI-I) Scales (NIMH, 1985a).
Description: The Clinical Global Impression - Improvement scale (CGI-I) is a 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. and rated as: 1. Very much improved; 2. Much improved; 3. Minimally improved; 4. No change; 5. Minimally worse; 6. Much worse; or 7. Much worse)
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aripiprazole Treatment of Conduct Disorder
Number analyzed (Participants) | 10
units on a scale | 2.1 (1.4)

ADVERSE EVENTS:
Time Frame: Subjects were enrolled for a 6 week study.
Description: Safety measures for extrapyramidal ADRs included the AIMS (NIMH, 1985b) for tardive dyskinesia Barnes Akathisia Scale (Barnes 1989) (BAS) and the Simpson-Angus Scale (SAS) for parkinsonian movements (Simpson and Angus 1970). The UKU (Lingjaerde et al 1987) was used for monitoring non-motor ADRs.
Groups:
- Aripiprazole in the Treatment of Conduct Disorder: The study was a 6-week open label study evaluating aripiprazole in the treatment of 12 male post-pubertal adolescents (13-17 years, Tanner Stage 4) diagnosed with conduct disorder (American Psychiatric Association 2000).
Arm/Group | Aripiprazole in the Treatment of Conduct Disorder
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 10/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aripiprazole in the Treatment of Conduct Disorder (N=10)
fatigue (General disorders) | 10 (29) — Increased fatigue, sleepiness-sedation, increased sleep duration, or decreased sleep duration
muscle rigidity (Nervous system disorders) | 4 — parkinsonian type symptoms of stiff muscles
tremor (Nervous system disorders) | 3 — tremor of extremities
akathisia (Nervous system disorders) | 5 — motor restlessness, increased pacing
Nausea/Vomiting (Gastrointestinal disorders) | 5
Increase perspiraton (Skin and subcutaneous tissue disorders) | 6
Head Aches (Nervous system disorders) | 9 — patient report on questionnaire
Weight Gain (Metabolism and nutrition disorders) | 4

LIMITATIONS AND CAVEATS:
12 subjects were recruited for this study but only 10 (83%) completed at least a week of data demonstrating the primary frustrations of the investigators in this study. Conduct disorder was a difficult diagnosis to recruit patients into this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2004-05-23): https://cdn.clinicaltrials.gov/large-docs/05/NCT00250705/Prot_000.pdf
  • Statistical Analysis Plan (2004-05-23): https://cdn.clinicaltrials.gov/large-docs/05/NCT00250705/SAP_001.pdf
  • Informed Consent Form (2004-05-23): https://cdn.clinicaltrials.gov/large-docs/05/NCT00250705/ICF_002.pdf